CLINICAL TRIAL: NCT03282526
Title: Volume Parameters Vs Flow Parameters In Assessment Of Reversibility In Stable Chronic Obstructive Pulmonary Disease Patients
Brief Title: Volume Parameters vs Flow Parameters in Assessment of Reversibility in Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Azza Bahaa El-Din Ali Mohamed, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: PFTs in COPD
Record Dates: First submitted 2017-08-26; First posted 2017-09-14 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Plethysmography, Whole Body; Spirometry

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole body plethysmography (Experimental)
  Interventions: Diagnostic Test: Whole body plethysmography
- spirometery (Active Comparator)
  Interventions: Diagnostic Test: Whole body plethysmography

INTERVENTIONS:
Diagnostic Test: Whole body plethysmography — Whole body plethysmography : measure lung volumes Spirometry : to assess severity of chronic obstructive pulmonary disease also reversibility testing
  Other Names: Spirometry; Plain chest radiograph

SUMMARY:
* Assess the differences between flow and volume responses after bronchodilator reversibility testing in patients over different clinical chronic obstructive pulmonary disease stages (GOLD stage I to GOLD stage IV).
* Study the Correlation between the bronchodilator response and the severity of the disease.

DETAILED DESCRIPTION:
chronic obstructive pulmonary disease is a common preventable and treatable disease characterized by persistent airflow limitation that is usually progressive. The diagnosis requires an evidence of obstructive pattern by spirometry measured before and after bronchodilators.

The degree of reversibility of airflow obstruction differs between patients, and does not predict the response to bronchodilator therapy. It can be seen in terms of forced vital capacity (FVC) or forced expiratory volume in the first second (FEV1),or Inspiratory capacity (IC) or residual volume (RV).

ELIGIBILITY:
Inclusion Criteria:

* Patients Clinical diagnosis of Chronic Obstructive Pulmonary Disease
* Must be able to do pulmonary function test
* Age more than 40 years
* Stable Chronic Obstructive Pulmonary Disease patients

Exclusion Criteria:

Any patients with a diagnosis of:

* Bronchial asthma
* Bronchiectasis
* Respiratory failure
* Decompensated core pulmonale
* Chronic Obstructive Pulmonary Disease combined with any other respiratory disease

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-09-30 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Assess the response pattern to inhaled short acting B2 agonist | twice per day one before inhaled short acting B2 agonist and one after 10 minutes from inhaled short acting B2 agonist for average of 2 year
  Assess the response pattern to inhaled short acting B2 agonist through measuring flow and volume parameters to define the differences between volumes responders and flow responders

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vogelmeier CF, Criner GJ, Martinez FJ, Anzueto A, Barnes PJ, Bourbeau J, Celli BR, Chen R, Decramer M, Fabbri LM, Frith P, Halpin DMG, Varela MVL, Nishimura M, Roche N, Rodriguez-Roisin R, Sin DD, Singh D, Stockley R, Vestbo J, Wedzicha JA, Agusti A. Erratum to "Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease 2017 Report: GOLD Executive Summary" [Arch Bronconeumol. 2017;53:128-49]. Arch Bronconeumol. 2017 Jul;53(7):411-412. doi: 10.1016/j.arbres.2017.06.001. No abstract available. English, Spanish. PMID 28668138
- [Result] "Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease 2017 Report: GOLD Executive Summary." Claus F. Vogelmeier, Gerard J. Criner, Fernando J. Martinez, Antonio Anzueto, Peter J. Barnes, Jean Bourbeau, Bartolome R. Celli, Rongchang Chen, Marc Decramer, Leonardo M. Fabbri, Peter Frith, David M.G. Halpin, M. Victorina Lopez Varela, Masaharu Nishimura, Nicolas Roche, Roberto Rodriguez-Roisin, Don D. Sin, Dave Singh, Robert Stockley, Jorgen Vestbo, Jadwiga A. Wedzicha and Alvar Agusti. Eur Respir J 2017; 49: 1700214. Eur Respir J. 2017 Jun 22;49(6):1750214. doi: 10.1183/13993003.50214-2017. Print 2017 Jun. No abstract available. PMID 28642306